CLINICAL TRIAL: NCT03588221
Title: Simplifying the WHO Protocol for Hand Hygiene: Three Steps and 15 Seconds - a Randomized Cross-over Trial
Brief Title: Simplifying the World Health Organization (WHO) Protocol for Hand Hygiene
Acronym: SIHAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 2018-01049;me18Tschudin-Sutter
Record Dates: First submitted 2018-07-03; First posted 2018-07-17 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Hand Hygiene

STUDY DESIGN:
Intervention Model Description: Randomized crossover trial, comparing the following four sets of hand hygiene measurements per participant:
  1. Six-step hand hygiene technique with an application time of 30 seconds
  2. Six-step hand hygiene technique with an application time of 15 seconds
  3. Three-step hand hygiene technique with an application time of 30 seconds
  4. Three-step hand hygiene technique with an application time of 15 seconds
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Six-step hand hygiene technique with application time of 30 (Other)
  Interventions: Procedure: four sets of hand hygiene measurements per participant
- Six-step hand hygiene technique with application time of 15 (Other)
  Interventions: Procedure: four sets of hand hygiene measurements per participant
- Three-step hand hygiene technique with application time of 3 (Other)
  Interventions: Procedure: four sets of hand hygiene measurements per participant
- Three-step hand hygiene technique with application time of 1 (Other)
  Interventions: Procedure: four sets of hand hygiene measurements per participant

INTERVENTIONS:
Procedure: four sets of hand hygiene measurements per participant — 1. Six-step hand hygiene technique with an application time of 30 seconds
  2. Six-step hand hygiene technique with an application time of 15 seconds
  3. Three-step hand hygiene technique with an application time of 30 seconds
  4. Three-step hand hygiene technique with an application time of 15 seconds

SUMMARY:
Non-inferiority in terms of reduction of bacterial counts will be investigated when combining the simpler three-step hand hygiene technique for the use of hand rub with a shorter application time of 15 seconds compared to the to the three steps technique with an application time of 30 seconds and the technique consisting in six steps.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (≥18 years)

Exclusion Criteria:

* skin disorders as determined by a dermatologist
* inability to follow procedures
* insufficient knowledge of the project language
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change of bacterial counts on hands pre and post hand hygiene measure | 30 minutes
  The log counts of bacteria detected on the dominant hand will be averaged separately for pre- and post values. Differences between pre- and post values, as well as in the mean logarithmic reduction in bacterial counts will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tschudin Sutter, PD MD, Principal Investigator — University Hospital Basel, CH-4031 Basel
Locations (1):
- Division of Infectious Diseases and Hospital Epidemiology, Basel, Switzerland